CLINICAL TRIAL: NCT07293520
Title: Improving Consent Experiences in Clinical Trials at Siteman Cancer Center
Brief Title: Improving Consent Experiences in Clinical Trials
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not receive funding
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202511065
Record Dates: First submitted 2025-12-05; First posted 2025-12-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Cancer
Keywords: Informed Consent; Key information; Research Ethics
MeSH Terms: conditions — Neoplasms | interventions — Electrophoresis, Polyacrylamide Gel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard consent forms (Active Comparator): The approved standard consent form will be used during the consent processes.
  Interventions: Behavioral: Standard Consent Form
- Standard consent forms with a visual key information (VKI) page (Experimental): The approved standard consent form with a VKI page will be used during the consent processes.
  Interventions: Behavioral: Standard Consent Form; Behavioral: Visual Key Information (VKI) page
- Research Team Members (Experimental): Members of the parent study's research team will complete the research team survey to assess opinions on consent process.
  Interventions: Behavioral: Standard Consent Form; Behavioral: Visual Key Information (VKI) page

INTERVENTIONS:
Behavioral: Standard Consent Form — The IRB-approved consent form will be used by research team staff during consenting process of participants for parent studies.
Behavioral: Visual Key Information (VKI) page — A VKI page will be designed for each parent study based on study materials and current consent document. The VKI will be implemented in the consent material for the study.
  Arms: Research Team Members; Standard consent forms with a visual key information (VKI) page

SUMMARY:
This is a study to evaluate the impact of evidence-based visual key information (VKI) pages on participant's experiences with informed consent for research, enrollment in high-accruing studies that choose to use VKIs as part of their consent process, and research team perceptions of the implementation potential of VKIs in studies. Unlike in previous pilots conducted at Siteman Cancer Center, this study will assess changes in outcomes before and after a VKI is implemented in a study consent process.

ELIGIBILITY:
Patient Eligibility Criteria:

* Patient must be 18 years or older
* Patients must be English-speaking
* Able to understand an IRB-approved written consent document
* Must go through the consent process for one of the parent studies

Research Team Eligibility Criteria:

* Member of a parent study research team
* Engaged in the study consent processes, including creating and reviewing consents or enrolling participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-11-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient's knowledge of consent | Time of consent completion for parent study (day 1)
  Knowledge of consent will be measured by patient's responses to 6-items on the patient consent experience survey. The 6-items are customized for each parent study and have three answers for patient to choose: true, false, and unsure. Responses will be reported via descriptive statistics and between group differences will be examined via chi-square tests.
Patient's anxiety about enrolling | Time of consent completion for parent study (day 1)
  Anxiety about enrolling will be captured by patient's answers to a single item on the patient consent experience survey adapted from the Amsterdam Preoperative Anxiety and Information Scale (APAIS). The item is measured by a 5-point Likert scale as follows: Not at all, A little, Somewhat, A lot, and Extremely. Responses be will scored as appropriate for the validated measure and between group differences will be examined via t-tests.

SECONDARY OUTCOMES:
Patient's trust in information | Time of consent completion for parent study (day 1)
  Patient's trust in information will be measured by a single-item on the patient consent experience survey adapted from the Health Information National Trends Survey (HINTS) from the National Cancer Institute. The item is a 5-point scale with answers as follows: Not at all, Slightly, Moderately, Very, and Extremely. Responses will be scored as appropriate for the validated measure and between group differences will be examined via t-tests.
Patient's perceptions of patient centered care | Time of consent completion for parent study (day 1)
  Perception of patient-centered care (PCC) will be measured by three items on the patient consent experience survey which are adapted from the Health Information National Trends Survey (HINTS) from the National Cancer Institute. The items are a 4-point scale as follows: Always, Usually, Sometimes, and Never. Responses will be scored as appropriate for the validated measure and between group differences will be examined via t-tests.
Parent study enrollment rates | Completion of enrollment (estimated total time is 9-13 months)
  Enrollment rates will be measured by total number of patients enrolled in each parent study. Responses will be reported via descriptive statistics and between group differences will be examined via t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Mary C Politi, PhD, Principal Investigator — Washington University in St. Louis School of Public Health

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu